CLINICAL TRIAL: NCT02253888
Title: An Open-label, Randomized, Single-dose, Two-way Crossover Bioequivalence Study Assessing Subjects Receiving Tipranavir 500 mg Stored at Controlled Temperature (Testproduct 30°C/70% RH) Compared With Tipranavir 500 mg Stored at Controlled Refrigerated Conditions (Reference Product 2-8°C), Orally Co-administered With Ritonavir 200 mg Under Fasting Conditions to Healthy Male and Female Volunteers
Brief Title: Bioequivalence Study of Tipranavir Stored at Controlled Temperature Compared With Tipranavir Stored at Controlled Refrigerated Conditions, Orally Co-administered With Ritonavir in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1182.93
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

ARMS (2):
- TPV/r - Room condition (Experimental)
  Interventions: Drug: TPV - Room condition; Drug: Ritonavir (RTV)
- TPV/r - Refrigerated conditions (Experimental)
  Interventions: Drug: TPV - Refrigerated conditions; Drug: Ritonavir (RTV)

INTERVENTIONS:
Drug: TPV - Room condition
  Arms: TPV/r - Room condition
Drug: TPV - Refrigerated conditions
  Arms: TPV/r - Refrigerated conditions
Drug: Ritonavir (RTV)

SUMMARY:
The objective of this trial was to establish the bioequivalence of Tipranavir (TPV) 250 mg self emulsifying drug delivery system (SEDDS) capsules that had been stored at a controlled temperature of 30°C and controlled relative humidity (RH) of 70% in comparison with TPV 250 mg SEDDS capsules stored at controlled refrigerated conditions between 2°C and 8°C

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females with a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG and clinical laboratory tests that have:

   * No findings that are abnormal or of clinical relevance
   * No evidence of a clinically relevant concomitant disease
   * Acceptable laboratory values that indicate adequate baseline organ function at time of screening. Laboratory values are considered acceptable if the severity is less than or equal to Grade 1, according to the AIDS Clinical Trials Group (ACTG) Division of Acquired Immunodeficiency Syndrome (of the National Institute of Allergy and Infectious Diseases / National Institutes of Health) (DAIDS) Grading Scale and within normal reference ranges for other laboratory parameters not defined by DAIDS. Participation of subjects with abnormal laboratory values greater than Grade 1 (e.g., Creatine phosphokinase (CPK), amylase, triglycerides) is subject to approval by the Boehringer Ingelheim Pharmaceuticals, Inc. (BIPI) clinical monitor
2. Age ≥18 and ≤60 years
3. Body mass index (BMI) ≥18.5 and ≤35.0 kg/m2
4. Signed and dated written informed consent before admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation concerning volunteers who are capable of understanding and giving informed consent
5. Willingness of subjects to abstain from ingesting the following foods and substances beginning 2 weeks before administration of any study medication and until the end of the study: grapefruit or grapefruit juice, red wine, Seville oranges, St. John's Wort and Milk Thistle
6. Willingness of subjects to abstain from use of alcohol within 72 hours before administration of study medication and to the end of the study
7. Willingness of subjects to abstain from the following substances within 72 hours before administration of study medication: garlic supplements and methylxanthine containing foods or drinks (including coffee, tea, cola, energy drinks, chocolate, etc.)

Exclusion Criteria:

1. Chronic gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy, cerebral cramps) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergies or hypersensitivity (including drug allergies) that are deemed relevant to the trial, as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within 1 month or less than 10 half-lives of the drug before administration of study drug or during the trial
8. Use of drugs that might reasonably influence the results of the trial (based on knowledge at the time of the protocol's preparation) within 10 days before administration of study drug or during the trial
9. Participation in another trial with an investigational drug within 30 days before administration of study drug or during the trial.
10. Smoker (more than 10 cigarettes per day, 3 cigars per day or 3 pipes per day)
11. Inability to refrain from smoking 24 hours before receiving study medication and on trial days when pharmacokinetic (PK) data are collected
12. High level of alcohol use (more than 60 grams per day)
13. Illicit drug use (i.e., positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
14. Veins unsuited for i.v. puncture on either arm (e.g., veins that are difficult to locate, access or puncture veins with a tendency to rupture during or after puncture)
15. Blood donation (more than 100 mL within 4 weeks before administration of study medication or during the trial)
16. History of any bleeding disorder or acute blood coagulation defect
17. Hypersensitivity to RTV or related antiretroviral drugs
18. Extreme physical activities (within 1 week before administration of study medication or during the trial)
19. Any laboratory value outside the reference range or >DAIDS Grade 1 that is of clinical relevance
20. Heart rate at screening of >90 bpm or <45 bpm
21. Seated systolic blood pressure either <95 mm Hg or >160 mm Hg
22. Any screening ECG value outside of the reference range of clinical relevance
23. Inability to adhere to dietary regimen of the study centre
24. For female subjects:

    * Pregnancy or planning to become pregnant within 60 days of study completion
    * Positive pregnancy test
    * Non-use of a barrier method of contraception for at least 3 months before participation in the study
    * Not willing or unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
    * Chronic use of oral contraception or hormone replacement containing ethinyl estradiol
    * Breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 hours extrapolated to infinity) | up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under concentration-time curve of the analyte in plasma over the time interval of 0 to time of last quantifiable data point) | up to 72 hours after drug administration
AUC0-72 (area under concentration-time curve of the analyte in plasma over the time interval t0h to t72h) | up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours after drug administration
λz (terminal rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz after an extravascular dose) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 11 days after last dose of drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 11 days after last dose of drug administration